CLINICAL TRIAL: NCT04354155
Title: COVID-19 Anticoagulation in Children - Thromboprophlaxis (COVAC-TP) Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: COVAC-TP
Record Dates: First submitted 2020-04-13; First posted 2020-04-21 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-03

CONDITIONS: Infection Viral; Thromboses, Venous; COVID-19
MeSH Terms: conditions — Virus Diseases; Venous Thrombosis; COVID-19 | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thromboprophylaxis (Experimental): Twice-daily low-dose enoxaparin thromboprophylaxis (starting dose, 0.5 mg/kg subcutaneously q12 hours, adjusted to achieve a 4 hour post-dose anti-factor Xa level of 0.20-0.49 anti-Xa U/mL)
  Interventions: Drug: Enoxaparin Prefilled Syringe [Lovenox]

INTERVENTIONS:
Drug: Enoxaparin Prefilled Syringe [Lovenox] — Twice-daily low-dose enoxaparin thromboprophylaxis (starting dose, 0.5 m/gkg subcutaneously q12 hours, adjusted to achieve a 4 hour post-dose anti-factor Xa level of 0.20-0.49 anti-Xa U/mL)

SUMMARY:
The purpose of this study is to evaluate the safety, dose-requirements, and exploratory efficacy of twice-daily subcutaneous enoxaparin as venous thromboembolism prophylaxis in children (birth to 18 years) hospitalized with signs and/or symptoms of SARS-CoV-2 infection (i.e., COVID-19).

ELIGIBILITY:
Inclusion Criteria:

1. Birth to <18 years of age; AND
2. Positive nucleic acid test for SARS-CoV-2 within the past 7 days; AND
3. Hospitalized, <72 hours post-admission; AND
4. One or more signs and/or symptoms of COVID-19 illness within the past 72 hours, as follows:

   1. Cough; OR
   2. Fever (oral temperature >100.4°F/38°C); OR
   3. Chest pain; OR
   4. Shortness of breath; OR
   5. Myalgia; OR
   6. Acute unexplained loss of smell or taste; OR
   7. New/increased supplemental oxygen requirement; OR
   8. Acute respiratory failure requiring non-invasive or invasive ventilation; OR
   9. Encephalitis.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Receiving therapeutic anticoagulation for treatment of a thromboembolic event diagnosed within the past 12 weeks; OR
2. Clinical-relevant bleeding (see criteria under Primary Outcome, below) within the past 72 hours; OR
3. Platelet count <50,000/µL within the past 24 hours; OR
4. Prothrombin time (PT) ≥2 seconds above the upper limit of age-appropriate local reference range within the past 24 hours; OR
5. Activated partial thromboplastin time (aPTT) ≥4 seconds above the upper limit of age-appropriate local reference range within the past 24 hours; OR
6. Fibrinogen level <75 mg/dL; OR
7. Severe renal impairment, as defined by estimated glomerular filtration rate (eGFR) <31 mL/min/ 1.73 m2, as calculated by the Schwartz formula; OR
8. Parent or legally authorized representative unwilling to provide informed consent for patient participation.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sochet, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (16):
- United States (16):
  - Children's of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Hemostasis and Thrombosis Center UC Davis, Sacramento, California
  - Rady Children's Hospital, San Diego, California
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Johns Hopkins Hospital and Children's Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Akron Children's Hospital, Akron, Ohio
  - Children's Hospital Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sochet AA, Sellers AR, Betensky M, Morrison JM, Ashour D, Fierstein JL, Amankwah EK, Bruzek S, Ignjatovic V, Goldenberg NA; COVID-19 Anticoagulation in Children-Thromboprophylaxis Trial Investigators. Immunothrombosis and plasma fibrinolytic function for pediatric COVID-19: a secondary analysis from the COVAC-TP trial. Blood Vessel Thromb Hemost. 2024 Nov 26;2(1):100038. doi: 10.1016/j.bvth.2024.100038. eCollection 2025 Feb. PMID 40766870
- [Derived] Sochet AA, Morrison JM, Jaffray J, Godiwala N, Wilson HP, Thornburg CD, Bhat RV, Zia A, Lawrence C, Kudchadkar SR, Hamblin F, Russell CJ, Streiff MB, Spyropoulos AC, Amankwah EK, Goldenberg NA; COVID-19 Anticoagulation in Children - Thromboprophylaxis (COVAC-TP) Trial Investigators. Enoxaparin Thromboprophylaxis in Children Hospitalized for COVID-19: A Phase 2 Trial. Pediatrics. 2022 Jul 1;150(1):e2022056726. doi: 10.1542/peds.2022-056726. PMID 35484817
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thromboprophylaxis
Started | 40
Completed | 38
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Did not meet criteria for study intervention | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data was not collected from 1 participant that withdrew and 1 participant who did not meet criteria for study intervention.
Arm/Group | Thromboprophylaxis
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 38
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Median Age (IQR) | 12.1 [1.3 to 17.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 12
  White | 16
  More than one race | 1
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Safety of In-hospital Thromboprophylaxis as Assessed by Number of Participants With ISTH-defined Clinically-relevant Bleeding Events During Hospitalization
Description: The safety of in-hospital thromboprophylaxis with twice-daily low-dose enoxaparin thromboprophylaxis will be measured by cumulative incidence (number of participants) of ISTH-defined clinically-relevant bleeding events during hospitalization. Clinically relevant bleeding episodes may include any of the following:
  1. fatal bleeding;
  2. clinically overt bleeding associated with a decline in hemoglobin of ≥2g/dL in a 24h period;
  3. retroperitoneal, pulmonary, or central nervous system bleeding;
  4. bleeding requiring surgical intervention in an operating suite;
  5. bleeding for which a blood product is administered (blood product administration not directly attributable to the patient's underlying condition);
  6. bleeding that requires medical or surgical intervention to restore hemostasis, other than in an operating suite.
Time Frame: Day 30
Population: There were 19 < 12 years of age and 19 >/= 12 years of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Thromboprophylaxis
Number analyzed (Participants) | 38
Participants | 0

2. Secondary Outcome: Median Twice-daily Enoxaparin Dose Required to Achieve 4-hour Post-dose Anti-factor Xa Between 0.20-0.49 U/mL
Description: The median twice-daily enoxaparin dose, as measured in mg/kg, required to achieve a 4-hour post-dose anti-factor Xa level of 0.20-0.49 anti-Xa U/mL in children hospitalized with COVID-19, and to compare dose-requirements by age group (<12 and those >12 years of age).
Time Frame: 4 hours post initial dose
Population: Analysis was done based on division of participants into two groups: < 12 years old and >/= 12 years old.
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Thromboprophylaxis
Number analyzed (Participants) | 38
mg/kg
  Children 12 years or older: number analyzed (Participants) | 19
  Children 12 years or older | 0.5 [0.46 to 0.52]
  Children less than 12 years: number analyzed (Participants) | 19
  Children less than 12 years | 0.52 [0.49 to 0.55]

3. Other Pre Specified Outcome: Efficacy of In-hospital Thromboprophylaxis as Measured by the Proportion of Serial D-dimer Levels
Description: To investigate, on a preliminary basis, the efficacy of in-hospital thromboprophylaxis with twice-daily enoxaparin in children hospitalized with COVID-19, as measured by the proportion of serial D-dimer levels obtained at standardized time points that are <2 times the upper limit of normal (<2x ULN) values for age.
Time Frame: Enrollment, Day 1, Day 2, and Day 3, 7, and 14 if still hospitalized
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Efficacy of In-hospital Thromboprophylaxis as Measured by Number of Participants With Confirmed HA-VTE
Description: To investigate, on a preliminary basis, the efficacy of in-hospital thromboprophylaxis with twice-daily enoxaparin in children hospitalized with COVID-19, as measured by number of participants with confirmed HA-VTE.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Thromboprophylaxis
Number analyzed (Participants) | 38
Participants | 2

ADVERSE EVENTS:
Time Frame: From enrollment through follow up, up to 30 days after enrollment.
Arm/Group | Thromboprophylaxis
All-Cause Mortality (participants affected / at risk) | 1/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04354155/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT04354155/SAP_001.pdf